CLINICAL TRIAL: NCT01833806
Title: A Phase IV Post Approval Clinical Study of ExAblate Treatment of Metastatic Bone Tumors for the Palliation of Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BM018; P110039/S2 (Other: FDA PMA Supplement)
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Bone Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ExAblate Test Arm (Experimental): Focused Ultrasound Surgery delivered by ExAblate MRgFUS
  Interventions: Device: ExAblate MRgFUS

INTERVENTIONS:
Device: ExAblate MRgFUS — Focused Ultrasound Ablation
  Other Names: Magnetic Resonance guided Focused Ultrasound Surgery

SUMMARY:
The study hypotheses is that the proportion of patients experiencing clinically significant pain relief will be at least 30% greater than the proportion experiencing worsening pain.

DETAILED DESCRIPTION:
As part of the PMA # P110039 review process and approval, InSightec was requested to conduct a post-approval study. Patients will be treated following the approved commercial treatment guidelines.

For this study, participating sites will use the ExAblate device for the administration of the ExAblate treatment. This study will be performed on either 1.5T or 3T MR scanners.

For this study, a total of 70 patients meeting the approved commercial guidelines will be enrolled and treated with the ExAblate system at from 7 to 10 sites. The proportion of responders is expected to be at least 30% greater than the proportion of subjects experiencing pain progression (i.e., 60% vs. 30%). Additionally, at the 3 month visit, an analysis of both the safety and efficacy profiles will be compared to the original PMA pivotal study group.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 and older
* Patients who are able and willing to give consent and able to attend all study visits
* Patients who are suffering from symptoms of bone metastases or multiple myeloma bone lesions:
* Patients who have received radiation without adequate relief from metastatic bone pain as determined by the patient and treating physician
* those for whom their treating physician would not prescribe radiation or additional radiation treatments
* patients who refuse additional radiation therapy.
* Patient with NRS (0-10 scale) pain score ≥ 4 irrespective of medication
* Targeted bone/tumor interface are ExAblate device accessible and are located in ribs, extremities (excluding joints), pelvis, shoulders and in the posterior aspects of the following spinal vertebra: Lumbar vertebra (L3 - L5), Sacral vertebra (S1 - S5)
* Targeted bone/tumor interface (most painful lesion) size up to 55 cm2 in surface area
* Patient whose targeted (treated) lesion is on bone and the interface between the bone and lesion is deeper than 10-mm from the skin.
* Targeted (treated) tumor clearly visible by non-contrast MRI, and ExAblate MRgFUS device accessible
* Able to communicate sensations during the ExAblate treatment
* Patients on ongoing chemotherapy regimen at the time of eligibility:

  1. with same chemotherapy regime (as documented from patient medical dossier), And
  2. Worst pain NRS still ≥ 4 And
  3. do NOT plan to initiate a new chemotherapy for pain palliation should be eligible for the study.

Note: Planned multiple courses of chemotherapy are not considered New Chemotherapy.

* No radiation therapy to targeted (most painful) lesion in the past two weeks Bisphosphonate intake should remain stable throughout the study duration.
* Patients will have from 1 to 5 painful lesions and only the most painful lesion will be treated.
* Patients with persistent distinguishable pain associated with 1 site to be treated (if patient has pain from additional sites, the pain from the additional sites must be evaluated as being less intense by at least 2 points on the NRS compared to the site to be treated).

Exclusion Criteria:

* Patients who either
* Need surgical stabilization of the affected bony structure (>7 fracture risk score, see Section 7.4) OR
* Targeted tumor is at an impending fracture site (>7 on fracture risk score, see Section 7.4).

OR

* Patients with surgical stabilization of tumor site with metallic hardware
* More than 5 painful lesions, or more than 1 requiring immediate localized treatment
* Targeted (treated) tumor is in the skull
* Patients on dialysis
* Patients with life expectancy < 3-Months
* Patients with an acute medical condition (e.g., pneumonia, sepsis) that is expected to hinder them from completing this study.
* Patients with unstable cardiac status including:
* Unstable angina pectoris on medication
* Patients with documented myocardial infarction within six months of protocol entry
* Congestive heart failure requiring medication (other than diuretic)
* Patients on anti-arrhythmic drugs
* Severe hypertension (diastolic BP > 100 on medication)
* Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
* Patients with an active infection or severe hematological, neurological, or other uncontrolled disease.
* Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease
* KPS Score < 60 (See "Definitions" below)
* Severe cerebrovascular disease (multiple CVA or CVA within 6 months)
* Individuals who are not able or willing to tolerate the required prolonged stationary position during treatment (approximately 2 hrs.)
* Target (treated) tumor is less then 1cm from nerve bundles, bowels or bladder.
* Are participating or have participated in another clinical trial in the last 30 days
* Patients initiating a new chemotherapy regime for pain purposes only, or radiation (for the targeted most painful lesion) within the last 2 weeks Note: Planned multiple courses of chemotherapy are not considered New Chemotherapy.
* Patients unable to communicate with the investigator and staff.
* Patients with persistent undistinguishable pain (pain source unidentifiable of the targeted lesion)
* Patient whose bone-lesion interface is < 10-mm from the skin
* Targeted (most painful) tumor NOT visible by non-contrast MRI,
* Targeted (most painful) tumor Not accessible to ExAblate
* The targeted tumor is less than 2 points more painful compared to other painful lesions on the site specific NRS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-09; Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - City of Hope, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - Mayo Clinic, Rochester, Minnesota
  - Weill Cornell Medical Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson, Houston, Texas
  - University of Virginia, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ExAblate Test Arm
Started | 32
Completed | 23
Not Completed | 9
Not completed — Alternative treatment | 2
Not completed — Death | 5
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | ExAblate Test Arm
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26
  Hispanic | 2
  Black | 1
  Asian | 3
Region of Enrollment [Number; unit: participants]
  United States | 32
Numerical Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Numerical Rating Scale (NRS) for pain is an 11 point scale ranging from 0 (no pain) to 10 (worst pain imaginable). Low scores (0) are better and high scales (10) are worse.
  units on a scale | 6.0 (1.71)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Responders
Description: The statistical hypothesis is that the proportion of responders will be significantly greater than the proportion of subjects experiencing pain progression (worsened pain or increased pain medications usage). Using the Numerical Rating Score (NRS) for pain (0 being no pain and 10 being worst imaginable pain), subjects were rated as a Responder or as having Pain Progression. A responder is defined as a subject with a reduction in NRS worst score from baseline of two (2) or more points, and no increase in pain medication use. Pain Progression was increased pain of two (2) or more points.
Time Frame: Three months post treatment
Population: The analysis was based on 31 treated subjects that completed at least one follow up visit; 23 out of 31 subjects were either Responders or had Pain Progression. Eight subjects reported no change in pain.
Measure: Count of Participants; unit: Participants
Arm/Group | ExAblate Test Arm
Number analyzed (Participants) | 31
Participants
  Responders | 18
  Pain Progression | 5
  No Change | 8
Statistical Analysis 1: Comparison: ExAblate Test Arm; The alternative hypothesis test was that the proportion of Responders would be greater than the proportion of subjects experiencing pain progression. This PAS was powered to enroll 70 subjects based on the pivotal trial proportion of 18:8 (Responders:Pain progression). The study was closed at an enrollment of 32 subjects; Test type: Superiority; p = 0.01, Binomial; Proportion Difference = 0.78, 95% CI 2-sided [0.58 to 0.98]

2. Other Pre Specified Outcome: Numerical Rating Scale (NRS) for Pain Score
Description: Patient pain intensity on an 11-point Numerical Rating Scale from 0 to 10 in which 0 is no pain and 10 is the worst pain you can imagine. The NRS was administered pre-treatment and post-treatment. The trajectory of change was presented graphically.
Time Frame: Three months post treatment
Population: There were 31 subjects treated that provided a baseline score and a final follow-up score.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ExAblate Test Arm
Number analyzed (Participants) | 31
score on a scale
  Baseline | 5.9 [5.28 to 6.43]
  1 Month Visit | 3.8 [2.93 to 4.65]
  2 Month Visit | 3.5 [2.56 to 4.54]
  3 Month Visit | 3.5 [2.31 to 4.66]

3. Other Pre Specified Outcome: Quality of Life (QOL) as Measured by Change in Brief Pain Inventory - Interference (BPI) From Baseline
Description: The BPI-QOL questionnaire is designed to show the severity and interference of pain in the lives of patients. This is a 7-item questionnaire that asks respondents the extent to which pain interferes with their general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life using a 0-10 numerical rating scale in which 0 represents 'does not interfere' and 10 indicates 'completely interferes'. Responses to the 7 items are averaged to form the pain interference scale score. Thus, the minimum possible is 0 and the maximum possible is 10 points. Lower scores are better, showing less interference in daily activities while higher scores show more interference and hence worse outcomes.
Time Frame: Baseline, 1 Month post treatment, 2 Month post treatment, 3 Month post treatment.
Population: One out of the 31 treated subjects did not complete the Baseline QoL (pain interference assessment and could not be included in the QoL analysis).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ExAblate Test Arm
Number analyzed (Participants) | 30
score on a scale
  Baseline | 5.0 [4.24 to 5.78]
  1 Month Visit | 3.4 [2.43 to 4.30]
  2 Month Visit | 3.2 [2.13 to 4.17]
  3 Month Visit | 3.1 [2.08 to 4.05]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 3 months following intervention.
Description: All device or procedure related adverse events were collected
Arm/Group | ExAblate Test Arm
All-Cause Mortality (participants affected / at risk) | 5/32
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 6/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ExAblate Test Arm (N=32)
Hypotension (Vascular disorders) | 1 (1) — While in post-procedure recovery the subject became hypotensive with a systolic pressure in the 70s. He was feeling well later that day. The even resolved within 3 days.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ExAblate Test Arm (N=32)
Sonication Pain (Surgical and medical procedures) | 2 (2)
Skin burn (Skin and subcutaneous tissue disorders) | 1 (1)
Skin peeled (Skin and subcutaneous tissue disorders) | 1 (1)
Blistering (Skin and subcutaneous tissue disorders) | 1 (1)
Sore lip (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT01833806/Prot_SAP_000.pdf